CLINICAL TRIAL: NCT06566339
Title: Robotically Assisted Anterior Eye Examinations for Acute Eye Care
Brief Title: Robotic OCT for ER Anterior Eye Exams
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00115313
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Develop and Test Robotically Assisted Imaging System for the Front of the Eye

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental: Imaging patients (Experimental): Participants eyes will be imaged with a Robotically aligned eye imaging system to help eye care through the emergency department
  Interventions: Device: Robotically Aligned Eye Imaging System
- Standard of care exam (No Intervention): ED providers' standard of care exam

INTERVENTIONS:
Device: Robotically Aligned Eye Imaging System — Robotically Aligned Eye Imaging System is a non-contact, micrometer scale imaging technique that provides clinicians and researchers with high resolution in vivo images sufficient to visualize layered microanatomy in 3D. The study team will develop hardware systems and software algorithms necessary for acquiring ocular anterior segment images for those seeking eye care in emergency department settings.
  Other Names: Robot OCT
  Arms: Experimental: Imaging patients

SUMMARY:
The purpose of this study is to develop and test a robotically assisted imaging system for the front of the eye with a goal of helping eye care through the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age and older
* Presenting with ocular complaints potentially indicative of an anterior segment pathology (e.g., foreign body sensation, red eye, pain)

Exclusion Criteria:

* Hemodynamically unstable patients (e.g., undergoing active resuscitation efforts)
* Patients with potential penetrating trauma to the eye who may need immediate surgical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Day 1
  Sensitivity of the ED providers' 1. standard of care exam and 2. assessment of robotically acquired ocular imaging to detect referable ocular pathology in the study participants will be compared. The on-duty ophthalmologist exam will serve as the gold standard.
Specificity | Day 1
  Specificity of the ED providers' 1. standard of care exam and 2. assessment of robotically acquired ocular imaging to detect referable ocular pathology in the study participants will be compared. The on-duty ophthalmologist exam will serve as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Kuo, MD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No